CLINICAL TRIAL: NCT03906435
Title: Parental Perception of Child Vulnerability in the NICU and Development Outcomes: A Randomized Control Trial Preventative Intervention With Cognitive Behavioral Therapy
Brief Title: Preventing Vulnerable Child Syndrome in the NICU With Cognitive Behavioral Therapy (PreVNT Trial)
Acronym: PreVNT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Margaret Hoge, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU 072018-095
Record Dates: First submitted 2019-03-19; First posted 2019-04-08 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Premature Infant; Mental Health Issue (E.G., Depression, Psychosis, Personality Disorder, Substance Abuse); Development, Child; Parent-Child Relations
Keywords: Vulnerable Child Syndrome; Neonatal Intensive Care Unit; Cognitive Behavioral Therapy; Parental Perception of Child Vulnerability; Child Developmental Outcomes; Parent Mental Health
MeSH Terms: conditions — Premature Birth; Depression; Psychotic Disorders; Personality Disorders; Substance-Related Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This will be a non-blinded randomized control to assess the outcomes of infants and parents receiving either Cognitive Behavioral Therapy (CBT) sessions focusing on NICU trauma, emotional responses, and parent perceptions of child vulnerability (PPCV) versus standard of care without CBT sessions.
  English and/or Spanish speaking parents of infants born at 30.6 weeks gestational age (GA) or less who survive to 33 weeks GA will be eligible to participate in the study. Once enrolled, the mother (and father, if willing) will be randomized into a control group (standard NICU and follow up care information) versus the intervention group (standard NICU and follow up care information plus a total of 5 CBT sessions split between the NICU and outpatient clinic visits post discharge from NICU). The CBT sessions will be standardized with a manual. Scales used for assessment will be distributed at enrollment to the study and upon completion of the CBT sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (No Intervention): Standard of care information given by NICU staff and Follow up Clinic staff, including information about health care, diagnosis, medications, daily cares, anticipatory guidance, and discharge prep information.
- Intervention CBT Arm (Experimental): In addition to Standard of care information that the control arm receives, this arm will also receive 5 CBT sessions focusing on past NICU trauma, emotional coping, parental perceptions of child vulnerability, and helpful parenting and emotional coping skills.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The intervention group will receive standard NICU and follow up care information plus a total of 5 CBT sessions split between the NICU and outpatient clinic visits post discharge from NICU. The CBT sessions will address PPCV in parents and parenting skills to address this. The CBT sessions will be standardized with a manual for study investigators to follow during sessions, and made with Dr. Richard Shaw from Stanford University, who wrote the prior CBT manual for anxiety, depression, and PTSD for NICU parents. Study staff will be trained to give the standardized CBT sessions using the manual via pilot sessions. There will be 3 CBT sessions given in the Parkland NICU before discharge and then 2 in the THRIVE follow up clinic at Children's Medical Center after discharge from the NICU.
  Arms: Intervention CBT Arm

SUMMARY:
This study is being done to see if outcomes for both a premature infant's parents and the infant born prematurely who have spent time in the neonatal intensive care unit (NICU) can be improved through parent cognitive behavioral therapy (CBT) sessions.

DETAILED DESCRIPTION:
The NICU is a stressful experience for parents. This stress naturally affects parents in different ways, ranging from feelings of depression, anxiety, or post traumatic stress disorder (PTSD). While these feelings are very common in parents of NICU children, they can also impact the ways parents perceive their infants, which leads to alterations of parenting styles and exposure to developmental activities for growing infants. This phenomenon is well described in the literature as Vulnerable Child Syndrome (VCS), or Parent Perceived Child Vulnerability (PPCV) to illness. Traumatic events from earlier experiences in the NICU usually cause PPCV to occur. Examples of traumatic events include feared death of the child, which lead to parent anxiety, depression, or emotional trauma. This altered perception of the child has been linked to worsened development outcomes for NICU children further out into childhood and also continued feelings of depression, anxiety, or fear in the parents and lack of confidence in their parenting abilities.

CBT sessions have been proven beneficial for NICU parents by decreasing feelings of depression, anxiety, and PTSD. However, there has not been research to see if CBT sessions are impactful for PPCV and the impacts it has on parent and child outcomes. Since literature suggests that depression, anxiety, and PTSD play an integral role in the development of PPCV and VCS, it could be assumed that CBT sessions should also be beneficial for PPCV and VCS. Therefore, this study will research if CBT sessions can improve parent-child interactions before and after discharge by helping parents to better understand their child's health and empower them with confidence in parenting skills. It will also evaluate if the effects of the CBT sessions will remain present and beneficial for parents' perceptions over time. With the results of this study, it will be evaluated if it is possible to improve the care for parents and children in the NICU as well as the long-term outcomes of parents and NICU children through CBT.

This will be a randomized control trial and will be conducted to assess the outcomes of infants and parents receiving either CBT sessions versus standard of care.

English and/or Spanish speaking parents of infants born at 30.6 weeks gestational age (GA) or less who survive to 33 weeks GA will be eligible to participate in the study. Families will be approached at 33 weeks GA to participate in the study. Once enrolled, the mother (and father, if willing to participate) will be randomized into a control group (standard NICU and follow up care information) versus the intervention group (standard NICU and follow up care information plus a total of 5 CBT sessions split between the NICU and outpatient clinic visits post discharge from NICU delivered either in person or virtually). The CBT sessions will address PPCV and VCS in parents and parenting skills to address preventing this. The CBT sessions will be standardized with a manual for study investigators to follow during sessions, and made with Dr. Richard Shaw from Stanford University, who wrote the prior CBT manual for anxiety, depression, and PTSD for NICU parents. Study staff will be trained to give the standardized CBT sessions using the manual via pilot sessions. There will be 3 CBT sessions given in the Parkland NICU before discharge and then 2 in the THRIVE follow up clinic at Children's Medical Center after discharge from the NICU. The investigators will look into the effects of in-person versus telehealth administration.

Scales used for assessment will be distributed at enrollment to the study and upon completion of the CBT sessions.

ELIGIBILITY:
Inclusion Criteria:

* Born at Parkland Hospital
* English or Spanish speaking mother +/- father
* ≤ 30.6 weeks gestation at birth
* Survival to 33 weeks gestation

Exclusion Criteria:

* Significant congenital anomalies
* Child Protective Services (CPS) involvement or foster care placement -- Prior enrollment in this PreVNT study for an older sibling.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
mean value score Vulnerable Baby Scale (VBSc) Score | difference in the mean value score of the VBSc scores of parents at baseline of the study (33 weeks post-menstrual age) versus at six to nine months of post-birth age
  Measures parental perceptions of child vulnerability. It has been used for parents with infants as young as 10-12 weeks of age up through 6 months to a year old. It is a 10 question scale, with each question scored on a five point likert scale (1-5). Score range is 10-50. Maximum score of 50 possible. A score of 27 or more was the median score for a sample of medically fragile neonates, and signifies relatively high perceptions of vulnerability. While a score of 23 was the median for a sample of healthy controls and thus reflect a more normal perception of vulnerability (Kerruish et al 2005). The higher the score, the higher the perception of child vulnerability.

SECONDARY OUTCOMES:
differences over time in subsets of Vulnerable Baby Scale (VBSc) scores | measurement differences over time between the total number of questions endorsed for each of the three different question subsets of VBSc of the parents at baseline of the study (33 weeks post-menstrual age) versus at six to nine months of post-birth age
  The VBSc can be broken down into subsets of questions addressing parent 1) thoughts: 2 questions of 10 scale questions, scored 0-2; 2) feelings: 3 questions of 10 scale questions, scored 0-3; and 3) actions/behaviors: 5 questions out of 10 scale questions, scored 0-5. This quantifies the amounts of subsets of the scale that the parent endorses. Higher numbers are markers of more and worse perceptions of child vulnerability in each category of thought, feeling, and action/behavior.
Correlation between changes over time in Vulnerable Baby Scale (VBSc) vs. Vulnerable Child Scale (VCSc) scores | measurement differences of scores from baseline of the study (33 weeks post-menstrual age) versus at six to nine months of post-birth age
  The VCSc is the most frequently and widely used scale to measure parent perceptions of vulnerability and Vulnerable Child Syndrome (VCS). It was modified by the author from the original 12 question scale to an 8 question scale. The modified scale has higher internal validity and consistency (Forsyth et al 1996). This scale was intended for and has been used for children aged mostly from 6 months to 8 years of age or older. Each question is scored on a four point likert scale (0-3). A total score of 0 to 24 is possible, the higher the score the more perceptions of vulnerability. A score of greater than 10 signifies high perceptions of vulnerability. See above for VBSc description.
differences over time in parent depression scores measured with Beck Depression Inventory Scale- 2nd edition. | measure differences of the scale's total score between timepoints at baseline of the study (33 weeks post-menstrual age) versus at six to nine months of post-birth age
  Beck Depression Inventory - 2nd Edition: This will be used to measure parent depression scores, which can be associated with development of VCS. This will be used as a secondary outcome in change over time throughout the study. This is a 21 item questionnaire, measured on a four point likert scale (0-3). A score of greater than 14 signifies depression, with higher scores representing more severe levels of depression. Scores of 0-13= No depression; 14-19= mild; 20-28= moderate; 29-63= severe.
child length of stay in the Parkland NICU (number of days) from birth to discharge from NICU, not including readmissions once first discharge has been accomplished. | Days will be counted that are spent in the NICU starting from the day of birth of the child which is the admission day to the NICU until discharge day that is documented from Parkland NICU, through study completion, an average of 1 year.
  child length of stay in the Parkland NICU (number of days) from birth to discharge from NICU, not including readmissions once first discharge has been accomplished. Scored in number of total days in the NICU (0 to infinite number). The higher the number, the more lengthy the NICU stay.
Child medical system usage score: number of non-well child or follow up visits/encounters until the last follow-up visit at 6-9 months averaged over the amount of months | from discharge from Parkland NICU until completion of the study at 6-9 months age
  The electronic medical record will be evaluated for how many total sick visits or hospital admissions are documented each month post discharge at Children's Medical Center and any associated hospitals that share medical records on the electronic medical record. The total number of encounters will be averaged over the amount of months from NICU discharge until the end of the study. Routine health checks will not be included in this number. A higher number will signify higher health care system usage.
differences over time in parent anxiety scores measured with Beck Anxiety Inventory Scale | measure differences of the scale's total score between timepoints at baseline of the study (33 weeks post-menstrual age) versus at six to nine months of post-birth age
  Beck Anxiety Inventory: This will be used to measure parent anxiety scores, which can be associated with development of VCS. This will be used as a secondary outcome for change over time throughout the study. This is a 21 item questionnaire, measured on a four point likert scale (0-3). Possible scores range from 0-36. A score of greater than 7 suggests anxiety. Scores of 8-15= mild; 16-25= moderate; 26-36= severe.
The Capute Scales: Cognitive Adaptive Test/Clinical Linguistic and Auditory Milestones Scale (CAT/CLAMS) | It will be administered at 6 months of age for all children enrolled in both study groups
  This is a neurodevelopmental tool used for children up through age 3 years old for cognitive assessment of infants and toddlers. It provides quantitative developmental quotients (DQ) for non-language visual motor (CAT DQ) and language (CLAMS DQ) abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret K Hoge, MD, Principal Investigator — UT Southwestern Medical Center Dallas; Roy Heyne, MD, Study Director — UT Southwestern Medical Center Dallas; Richard J Shaw, MD, Study Director — Stanford University
Locations (1):
- Parkland Health & Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
There will be a data sharing agreement signed between all parties and institutions to agree to share data safely and confidentially if sharing is necessary. The data shared will be de-identified for the purposes of data analysis and result interpretation.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: upon start of study to completion of study and manuscript submission.

REFERENCES:
- [Background] Kerruish NJ, Settle K, Campbell-Stokes P, Taylor BJ. Vulnerable Baby Scale: development and piloting of a questionnaire to measure maternal perceptions of their baby's vulnerability. J Paediatr Child Health. 2005 Aug;41(8):419-23. doi: 10.1111/j.1440-1754.2005.00658.x. PMID 16101975
- [Background] Forsyth BW, Horwitz SM, Leventhal JM, Burger J, Leaf PJ. The child vulnerability scale: an instrument to measure parental perceptions of child vulnerability. J Pediatr Psychol. 1996 Feb;21(1):89-101. doi: 10.1093/jpepsy/21.1.89. PMID 8820075
- [Derived] Hoge MK, Heyne E, Brown S, Heyne R, Shaw RJ, Chalak L. Reduction of neonatal intensive care unit (NICU) parental perceptions of child vulnerability and risk of vulnerable child syndrome utilizing cognitive behavioral therapy: randomized controlled trial. Pediatr Res. 2025 May 15. doi: 10.1038/s41390-025-04094-x. Online ahead of print. PMID 40374965